CLINICAL TRIAL: NCT05527301
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy and Safety of HEM1036 in Subjects With Low Anterior Resection Syndrome (LARS)
Brief Title: HEM1036 Phase 2 Study in Low Anterior Resection Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HEM Pharma Inc. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HEM_HEM1036_01
Record Dates: First submitted 2022-08-08; First posted 2022-09-02 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: LARS - Low Anterior Resection Syndrome
Keywords: LARS - Low Anterior Resection Syndrome; Probiotics; Colorectal Cancer
MeSH Terms: conditions — Low Anterior Resection Syndrome; Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEM1036 (Lactobacillus fermentum) (Experimental): Daily dose of 1 × 10^10 colony-forming units divided in 2 equal doses as a powder for BID oral administration
  Interventions: Drug: Lactobacillus Fermentum
- Placebo (Placebo Comparator): 2g Powder for BID oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lactobacillus Fermentum — Lactobacillus Fermentum
  Other Names: HEM1036
  Arms: HEM1036 (Lactobacillus fermentum)
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Double-blind, randomized, placebo controlled phase 2 study to explore the efficacy and safety of HEM1036 in the treatment of subjects with LARS

DETAILED DESCRIPTION:
The study will be conducted as a double-blind, randomized, placebo controlled phase 2 study to explore the efficacy and safety of HEM1036 in the treatment of subjects with LARS. Subjects will be males and females ≥18 and ≤75 years of age with LARS. Subjects must have a LARS score of >20 at the Screening Visit after sphincter preserving rectal resection surgery for the curative treatment of diagnosed rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects ≥18 and ≤75 years old.
2. Diagnosed with rectal cancer and undergone sphincter preserving rectal resection surgery.
3. Completed curative treatment (rectal resection, systemic chemotherapy, hormonal therapy, immunotherapy, biologic therapy, radiotherapy, and stomy repairment) ≥6 months prior to Screening.
4. Current LARS with a LARS score >20 at Screening.
5. An Eastern Cooperative Oncology Group score 0 or 1 at Screening.
6. No evidence of anastomotic leakage or severe stenosis.
7. Capable of returning to study site for all study visits according to requirement of protocol and willing to comply with the policy, procedure, and restriction of the study.
8. Capable of actively communicating with the investigator/study personnel and completing the study related documents.
9. Body mass index is at least 18 kg/m2 but no more than 35 kg/m2.

Exclusion Criteria:

1. History of: Abdominoperineal resection surgery, Hartmann operation, colostomy, Transanal irrigation therapy for LARS within 2 weeks prior to Screening, Secondary operation with stoma, etc.
2. Not completed stomy repairment done at rectal resection surgery.
3. History of allergic or adverse responses to IP or Milk, yeast, soy.
4. On systemic chemotherapy, hormonal therapy, immunotherapy, biologic therapy, or radiotherapy at the time of Screening.
5. Any antibiotic use within 4 weeks before the first dose of the IP.
6. Is currently participating or has participated in another study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of the IP.
7. Tested positive for HIV antigen, Hepatitis B, C at screening
8. Past or current alcohol or drug abuse history

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Low Anterior Resection Syndrome score from Baseline to 8 weeks | Baseline to 8 weeks
  * Higher score means worse outcome
  * We will assess the change of LARS score at 8 weeks frome baseline. The change of LARS score of two treatment groups will be compared.

SECONDARY OUTCOMES:
Change in QoL(Quality of Life) score from Baseline to 8 weeks | Baseline to 8 weeks
  Score 0-100(higher score means better outcome)
Change in fecal microbiota composition assessed by alpha-diversity and differential abundance analysis | Baseline to 4, 8 weeks
Change of fecal metabolites assessed by fecal analysis | Baseline to 4, 8 weeks
  Change of metabolites (including Total short-chain fatty acids, acetate, butyrate,propionate, lactate, bile acids in fecal samples) assessed by fecal analysis and all parameters will be presented as umol/g

IPD SHARING:
Plan to Share IPD: No